CLINICAL TRIAL: NCT01895530
Title: Impact of Probiotics in Modulation of Intestinal Microbiota of Patients Undergoing a Resection Colonic
Brief Title: Impact of Probiotics in Modulation of Intestinal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Isabel Toulson Davisson Correia (Other)
Responsible Party: Sponsor-Investigator, Maria Isabel Toulson Davisson Correia, PhD., Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ETIC 0391.0.203.000-09
Record Dates: First submitted 2013-06-30; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: Probiotics; colorectal cancer; postoperative infection; immune function; bacterial translocation; gastrointestinal surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Conventional treatment with no probiotic supplementation
- Probiotic group (Experimental): The patients received one oral lyophilized yeast capsule, each of which contains 100 mg (0,5 x 109 cfu/g) of Saccharomyces boulardii (Merck S.A., Biocodex, Beauvais, French), once a day. The treatment started at least seven days before surgery and stopped on the operation day.
  Interventions: Dietary Supplement: Saccharomyces boulardii

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii — The patients received one oral lyophilized yeast capsule, each of which contains 100 mg (0,5 x 109 cfu/g) of Saccharomyces boulardii (Merck S.A., Biocodex, Beauvais, French), once a day. The treatment started at least seven days before surgery and stopped on the operation day.
  Arms: Probiotic group

SUMMARY:
The investigators would study about impact of the administration of probiotics in the intestinal mucosa of patients undergoing resection colic, by evaluating cytokine profile by quantitative real time PCR. The investigators believe that patients who use probiotic preoperative would provide cytokine profile less inflammatory than those of the control group.

DETAILED DESCRIPTION:
Samples of colorectal cancer-free mucosa derived from patients who underwent surgical resection were investigated. Quantitative real-time polymerase chain reaction (RT-qPCR) was used to determine expression levels of the following genes: IL10, IL1B, IL23A, TNF, IL12B, INFG, IL17A.

ELIGIBILITY:
Inclusion Criteria:

* if he or she were older than 18 years
* intended to undergo elective CRC resection at UFMG Hospital

Exclusion Criteria:

* Patients were excluded if they were not able to receive the probiotics seven days before the operation
* if colon resection was not performed due to changes in operation strategy, or if they discontinued probiotic use on their own or
* if they removed their consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference in gene expression of citokynes | 15 days
  Colonic mucosal specimens were analyzed to determine the mucosal expression proﬁles of IL1B, IL12B, IL10, IL23A, INFG, IL17A and TNF.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Postoperative complications assessed up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabel TD Correia, PhD, Study Director — Federal University of Minas Gerais
Locations (1):
- UFMG Hospital, Belo Horizonte, Minas Gerais, Brazil